CLINICAL TRIAL: NCT00146822
Title: ENDOTAK RELIANCE G Evaluation of Handling and Electrical Performance Study
Brief Title: REFLEx Study (ENDOTAK RELIANCE G Evaluation of Handling and Electrical Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CR-CA-022504-L
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

INTERVENTIONS:
Device: ENDOTAK RELIANCE G lead

SUMMARY:
The REFLEx Study will evaluate if ENDOTAK RELIANCE G defibrillation leads with GORE ePTFE-covered coils are as good as or better than other comparative commercially available defibrillation leads with respect to electrical performance and termination efficacy in spontaneous tachyarrhythmic episodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current ICD or CRT-D indications
* Patients who are going to be implanted with one of the aforementioned ICD or CRT-D devices
* Patients who are going to be implanted with active-fixation, dual-coil, endocardial defibrillation leads with compatible connectors (i.e., ENDOTAK RELIANCE G or study-comparative ICD leads)
* Patients who sign and date a Patient Informed Consent form prior to device implant
* Patients who remain in the clinical care of the enrolling physician in approved centers
* Patients who are at least 18 years old

Exclusion Criteria:

* Patients who have a preexisting transvenous lead system that is not completely explanted
* Patients who are hypersensitive to a single dose of approximately 1.0 mg of dexamethasone acetate
* Patients who are expected to receive a heart transplant during the duration of the study
* Patients whose estimated life expectancy is less than 12 months due to other medical conditions
* Patients who currently have or who are likely to receive a tricuspid valve prosthesis
* Patients who are likely to have an open-chest surgery in the next three months
* Patients who are currently enrolled in another investigational study that would directly impact the treatment or outcome of the REFLEx study.
* Patients who are mentally incompetent and cannot sign a Patient Informed Consent form or comply with the study
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500
Dates: Start 2004-02; Study Completion 2006-03

PRIMARY OUTCOMES:
Lead electrical properties
First shock conversion success rate for spontaneous fast ventricular tachycardia or ventricular fibrillation

SECONDARY OUTCOMES:
Lead handling characteristics
Lead migration/dislodgment rates
Characterize the current ICD/CRT-D population
Effects of ischemia and revascularization and previous lead extraction on the lead's electrical performance

CONTACTS AND LOCATIONS:
Overall Officials: Randolph Cooper, MD, Principal Investigator — Wake Heart Associates